CLINICAL TRIAL: NCT06184295
Title: Robotic Balance Training to Improve Postural Control and Balance Post-Traumatic Brain
Brief Title: Robotic Balance Training to Improve Postural Control and Balance Post-Traumatic Brain Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Kiran Karunakaran, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-1229-23
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- TBI - Intervention Group (Experimental): The participants will receive 10 customized robotic balance training sessions to improve balance using the Hunova robotic device. Each session will last for up to 1.5 hours. The training may include standing or sitting on the robotic balance platform and performing the following tasks: maintaining balance when the platform becomes unstable or moving in various directions, or in an inclination; these tasks may be performed as instructed with eyes open or eyes closed condition; move in different directions to reach targets with my hands; stand on one leg or heel to toe and maintain balance; perform head or torso rotation while standing or sitting. All training will be performed with an overhead harness and a spotter will be present at all times.
  Interventions: Device: TBI - Intervention Group
- TBI - Non Intervention Group (No Intervention): Participants will receive no intervention
- Participants without disability group (No Intervention): Participants will receive no intervention

INTERVENTIONS:
Device: TBI - Intervention Group — The participants will receive 10 customized robotic balance training sessions to improve balance using the Hunova robotic device. Each session will last for up to 1.5 hours. The training may include standing or sitting on the robotic balance platform and performing the following tasks: maintaining balance when the platform becomes unstable or moving in various directions, or in an inclination; these tasks may be performed as instructed with eyes open or eyes closed condition; move in different directions to reach targets with my hands; stand on one leg or heel to toe and maintain balance; perform head or torso rotation while standing or sitting. All training will be performed with an overhead harness and a spotter will be present at all times.
  Arms: TBI - Intervention Group

SUMMARY:
The purpose of this study is to assess a balance training program to see if it can be helpful to improve balance and avoid falls in people who have had traumatic brain injuries (TBIs).

The study will involve three groups of research subjects: 1) TBI-intervention group, 2) TBI- non-intervention group and 3) the participants without disability group.

The TBI intervention Group will participate in 10 robotic balance training sessions. Data will collected pre and post-training.

TBI- non-intervention group will not receive any training. They will participate in two data collection sessions which are about 5 weeks apart.

The participants without disability group will not receive any training. They will participate in one data collection session.

ELIGIBILITY:
Participants with TBI:

Inclusion Criteria:

* Be between the ages of 18 and 65.
* Have been diagnosed with a TBI by a physician and be at least 6 months post injury and not more than 5 years post injury.
* Have been medically stable for 3 months prior to the most recent TBI.
* Not plan to make any drastic changes to medications (as determined by study staff) for at least 4 weeks.
* Be able to stand unsupported for 5 minutes.
* Be willing and able to give informed consent.
* Be able and willing to comply with study procedures, verbal instructions, and follow-up requirements.

Exclusion Criteria:

* Weight above 300 lbs.
* Have severe cardiac disease such as heart attack or moderate or severe congestive heart failure.
* Have a pre-existing condition resulting in significant disruption in alignment or function of the lower limb during standing.
* Have additional medical conditions that affect the bones, muscles or nerves that would interfere with the balance.
* Have any previously diagnosed history of balance problems prior to TBI.
* Have fluctuating blood pressure.
* Be on any medication that may affect balance, strength, or muscle coordination (e.g. Botox).
* Be currently enrolled in another research study that is likely to affect participation in this research study.
* Have seizure disorder.

Participants without a disability:

Inclusion Criteria:

* Be between the ages of 18 and 65.
* Not plan to make any drastic changes to medications for at least 4 weeks.
* Not have an orthopedic, cognitive or neuromuscular disease.
* Be able to stand unsupported for 5 minutes.
* Be willing and able to give informed consent.
* Be able and willing to comply with study procedures, including follow-up requirements.

Exclusion Criteria:

* Weight above 300 lbs.
* Have a history of injury to my lower limbs in the past 90 days.
* Have severe cardiac disease such as heart attack or moderate or severe congestive heart failure.
* Have a pre-existing condition resulting in significant disruption in alignment or function of the lower limb during standing.
* Have any additional medical conditions that affect my bones, muscles, or nerves that would interfere with the movement or the ability to feel touch or pain.
* Have difficulty following or responding to commands that would limit the study participation.
* Be currently enrolled in another research study that is likely to affect participation in this research study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Assessment | 5 weeks
  A task performance test consisting of 14 items of increasing difficulty graded on a five-point ordinal scale of 0 to 4 (0 = subject is unable to perform task; 4 = subject is independent in performance of task) giving the best possible score of 56 for healthy balance.
Dynamic Gait Index | 5 weeks
  Dynamic Gait Index (DGI) is a measurement tool commonly used to assess dynamic balance, gait and risk for falls. It consists of a total of eight gait assessments which can be scored on a four-point ordinal scale, ranging from 0-3, where '0' indicates the lowest level of function and '3' the highest level of function, allowing for a total possible score of 24.
Timed Up and Go | 5 weeks
  It is a clinical test of functional gait abilities and dynamic balance. The participants will be asked to walk a distance of 3 meters from a seated position, turn around, walk back to the chair and sit back in the chair. The time taken to perform the task will be recorded using a stopwatch.
10 Meter walk test | 5 weeks
  Participants will be asked to walk about 12 meters. The time taken to walk 10 meters will be recorded.
Fall Efficacy Scale -International | 5 weeks
  This questionnaire is a widely accepted tool for the assessment of fear of falling and has excellent reliability and validity. It is a self-reported questionnaire that provides information on the level of concern about falls for a range of daily living activities. The original questionnaire contains 16 items and is scored on a four-point scale (1 = not very concerned to 4 = very concerned). Therefore the best possible value is 16 and the worst is 64.
Community Balance and Mobility Scale | 5 weeks
  Used to detect 'high level' balance and mobility deficits based on tasks commonly encountered in community environments. Composed of 13 challenging tasks (scaled from 0 = complete inability to perform task to 5 = most successful completion of item available).
Temporal- spatial characteristics | 5 weeks
  Participants will be asked to walk about 10 meters on a pressure mat. Pressure mat (ZenoMat, Protokinetics LLC) will be used to collect gait cycle times and step length, in order to determine inter- and intra-limb temporal and spatial characteristics.
Electromyography | 5 weeks
  surface Electromyography (EMG) wireless sensors will be used to measure the activation of tibialis anterior, soleus, vastus lateralis, rectus femoris, bicep femoris, and gastrocnemius.
Cortical activity | 5 weeks
  Cortical activity will be measured using NIRSport 2 (NIRX Medical Technologies, LLC ), an Functional Near Infrared Spectroscopy (fNIRS) system. NIRSport 2 is a portable, non-invasive optical imaging technique to measure the cerebral hemodynamic response.
Balance | 5 weeks
  Quantitative measures of static and dynamic balance will be assessed using the Hunova balance platform.

SECONDARY OUTCOMES:
community ambulation | 5 weeks
  Sensors will be provided to be worn in wrist, leg and waist to collect gait cycle times and step length during community ambulation of the participants between baseline and follow-up. The participants will also wear the sensor during testing walking and balancing tasks at baseline and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Karunakaran, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided